CLINICAL TRIAL: NCT00240565
Title: A Single Arm, Open-label, Multicentre, Phase II Study of Tositumomab and Iodine 131-Tositumomab in Subjects With Indolent Non-Hodgkin's Lymphoma Who Have Previously Received Rituximab.
Brief Title: Tositumomab And Iodine I 131-Tositumomab In Patients With Relapsed Indolent Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 393229/032
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2012-08-13 (Estimated); Status verified 2012-08

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: BEXXAR; non-Hodgkin's Lymphoma; tositumomab; I-131
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — tositumomab I-131

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Participants underwent two phases of treatment: an initial DD, followed by a therapeutic dose. The one-day DD comprised a 1 hr IV infusion of 450 mg unlabeled TST, followed by a 20 min IV infusion of 35 mg TST labeled with 185 MBq (5.0 mCi) of I 131. After 7 to 14 days, the one-day therapeutic dose comprised a second 1 hr IV infusion of 450 mg unlabeled TST, followed by a 20 min IV infusion of 35 mg TST labeled with I 131 with an administered activity (MBq or mCi) determined from the dosimetry calculation.
  Interventions: Drug: Tositumomab 450 mg; Drug: Tositumomab 35 mg

INTERVENTIONS:
Drug: Tositumomab 450 mg — Unlabeled TST
Drug: Tositumomab 35 mg — TST labeled with 185 megaBecqueral (mbq) of iodine 131

SUMMARY:
This study will further characterize the activity of Tositumomab and Iodine I 131-Tositumomab in patients with relapsed indolent non-Hodgkin's Lymphoma who have progressed following treatment with rituximab.

ELIGIBILITY:
Inclusion criteria:

* Patients must have evidence of persistent or progressive follicular grade, 1, 2 or 3 or marginal zone B-cell non-Hodgkin's lymphoma.
* Must have received at least two prior courses of systemic treatment including at least one treatment of rituximab (lymphoma must not have progressed during their most recent systemic chemotherapy treatment).
* Must have evidence that their lymphoma expresses CD20 antigen and have adequate renal and hepatic function.

Exclusion criteria:

* Received chemotherapy, radiation therapy, immunosuppressants or cytokine treatment within 4 weeks prior to study entry.
* Have active obstructive hydronephrosis.
* Had prior autologous hematopoietic stem cell transplant or any allogenic stem cell transplant.
* Have active infection requiring IV antibiotics.
* Have brain or leptomeningeal metastasis.
* Had previous allergic reaction to iodine, previously received radioimmunotherapy or are currently receiving approved or experimental anti-cancer drugs.
* Patients who are pregnant or breast feeding, have known HIV infection, or are Human anti-murine antibody (HAMA) positive.
* Other criteria will be evaluated at the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2004-04; Primary Completion 2007-02 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Response Rate | Week 26
  Responders are defined as participants with Complete Response (CR: disappearance of all clinical and radiological evidence of lymphoma), Clinical Complete Response (CCR: all criteria met for CR, except there is a residual nodal mass >15 millimeters), or Partial Response (PR: 50% reduction in the sum of the products of the longest perpendicular diameters of all measurable lesions with no new lesions). Response is based on objective evaluation, using the guidelines developed by The International Workshop to Standardize Response Criteria, independent of the investigator's evaluation.

SECONDARY OUTCOMES:
Complete response rate (CR) | From the start of treatment (Study Day 0, Baseline) until long-term follow-up (every 6 months until 5 years from the time of study entry)
  Investigator-assessed confirmed CR is defined as the disappearance of all clinical and radiological evidence of lymphoma. Response is based on objective evaluation, using the guidelines developed by The International Workshop to Standardize Response Criteria, independent of the investigator's evaluation.
Duration of response | 5 years
  Duration of response is defined as the time from the first documented response to the first documented disease progression. Response is based on objective evaluation, using the guidelines developed by The International Workshop to Standardize Response Criteria, independent of the investigator's evaluation. Disease progression is defined as a 50% increase in the sum of the products of the two perpendicular diameters of all measurable lesions, or the appearance of new lesions.
Progression-free survival (PFS) | 5 years or until death
  PFS is defined as the time interval between the date of the DD to the first date at which progressive disease (PD) or death is observed. PD is defined as a 50% increase in the sum of the products of two perpendicular diameters of all measurable lesions, or the appearance of new lesions. Participants with no evidence of PD were censored to the last date of contact; and those who died for any reason in the absense of PD were classified as having experienced PD on the date of death. For non-responders, duration of PFS was recorded as 0. Participants were censored if they withdrew without PD.
Adverse events | 5 years or until death
  An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. A serious adverse event (SAE) is any untoward medical occurrence that, at any dose results in death; is life-threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; is a congenital anomaly in a child from a parent who was exposed to treatment; or is an SAE based on medical or scientific judgement of the investigator.
Quality of Life | 5 Years
  Qualty of Life will be asessed utilizing several scales and questionnaires: FACT-G questionnaire was designed to measure multidimensional quality of life (QOL) in participants with cancer. FACT-LymThe FACT-Lym subscale questionnaire is a cancer-specific questionnaire designed to measure multidimensional QOL in participants with lymphoma.
Resource Utilization Assessment | Week 26
  The Resource Utilization Assessment questionnaires are used to assess the resource utilization of the participant and impacted associates (e.g., family members, caregivers) as well as costs involved to treat participants receiving TST and I 131 TST. As an assessment of general health, participants were asked to rate their activity level on average in the last 7 days on an 11-point scale: 0= exhausted in bed all day; 10=normal activity level.
Duration of Overall Survival | 5 years or until death
  Survival time is defined as the number of weeks from the first study medication administration to the date of death. In the absence of confirmation of death, survival time was censored to the last date the participant was known be alive. If the participant was alive at the time of analysis, then the survival time was censored at the date of last contact.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- Canada (8):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec

REFERENCES:
- [Derived] Olney HJ, Freeman MA, Stewart DA, Mangel JE, White DJ, Elia-Pacitti JO. Prolonged progression-free survival and preserved quality of life in the Canadian prospective study of tositumomab and iodine(131)-tositumomab for previously treated, rituximab-exposed, indolent non-Hodgkin lymphoma. Leuk Lymphoma. 2014 Dec;55(12):2754-60. doi: 10.3109/10428194.2014.894190. Epub 2014 Apr 3. PMID 24528219